CLINICAL TRIAL: NCT07164417
Title: Comparing Two Types of PRF Membranes in Management of Dehiscence Defect With Simultaneous Implant Placement in Posterior Mandible (Randomized Controlled Clinical Trial)
Brief Title: Two Types of PRF Membranes in Management of Dehiscence Defect in Posterior Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0936-06/2024
Record Dates: First submitted 2025-09-04; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Atrophic Mandible

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRF (Active Comparator)
  Interventions: Other: PRF membrane will be used with xenograft simultaneously with implant placement
- e-PRF (Experimental)
  Interventions: Other: e-PRF membrane will be used with xenograft simultaneously with implant placement.

INTERVENTIONS:
Other: e-PRF membrane will be used with xenograft simultaneously with implant placement. — Peripheral blood is collected in plain tubes and centrifuged (700-2000 g, 8 min) to separate plasma from red cells. The first 2-4 mL of platelet-poor plasma (PPP) is withdrawn and heated at 75 °C for 10 minutes to form albumin gel, then cooled for 1-2 minutes. Meanwhile, the remaining blood fractions (buffy coat, liquid PRF, red cells) are kept cooled to prevent premature clotting.
  Arms: e-PRF
Other: PRF membrane will be used with xenograft simultaneously with implant placement — Peripheral blood is collected in 9-10 mL additive-free tubes and centrifuged horizontally at 700-2000 g for 8 minutes.
  Arms: PRF

SUMMARY:
Background: Placement of implants in an atrophic posterior ridge is a challenge for so many clinicians. The success of dental implants depends on the volume of alveolar bone available to provide stability. Bone grafting using xenograft with PRF and e-PRF as a membrane has shown promising results in both bone healing and defect reconstruction. Aim of the study: to evaluate the effect of Platelet-rich fibrin (PRF) and Extended Platelet-rich fibrin (e-PRF) as a membrane with xenograft to increase the width of ridge in posterior mandible with simultaneous implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patient with one or more missing posterior mandibular teeth.
* Patient with atrophic posterior mandible with residual ridge width in the range of 4 to 6mm.
* Patient with good oral hygiene and acceptable inter-arch space less than or equal to the restoration

Exclusion Criteria:

* The patient underwent alveolar ridge reconstruction in the same area.
* Patients with immune diseases, uncontrolled hypertension, and uncontrolled diabetes.
* Patient with any pathological condition at the site of surgery.
* Heavy smoker, alcohol abuse, parafunctional habits.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change in implant stability | baseline and 6 months
  Osstell device will be used to measure the implant stability, primary stability Just after implant placement, and secondary stability 6 months from the time of implant placement. The measured values will be recorded in ISQ from 1 to 100, Implant stability is directly proportional to ISQ value

SECONDARY OUTCOMES:
change in pain scores | uo to 7 days
  Visual Analogue Scale (VAS) will be used to assess pain for 7 days postoperatively using a 10-point (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Change in edema scores | up to 7 days
  Assessment of edema will be done immediately, post-operative on the 2nd, 3rd, and 7th days as follows:
  no inflammation= none intraoral swelling confined to the surgical field = mild extraoral swelling in the surgical zone= moderate extraoral swelling spreading beyond the surgical zone= intense
change in bone width gain | baseline and 6 months
  CBCT will be used
change in bone density | baseline and 6 months
  CBCt will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt

IPD SHARING:
Plan to Share IPD: No